CLINICAL TRIAL: NCT06615232
Title: The Impact of Vaginal Washing on Cervical Inflammation: A Randomized Controlled Trial
Brief Title: The Impact of Vaginal Washing on Cervical Inflammation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle Sabo, Acting Assistant Professor: School of Medicine, Allergy and Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00021251; R01HD115465 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Reproductive Behavior
Keywords: sex work; hiv; vaginal washing; cervicovaginal inflammation; mucosal barrier disruption
MeSH Terms: conditions — Reproductive Behavior; Sex Work; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Women will be randomized in groups of 20 to either the vaginal washing cessation intervention or control (no intervention) arm. Women randomized to the intervention arm will attend 3 small group sessions over the course of a month focused on sexual health education and vaginal washing cessation. Women in both groups will be asked to provide samples (vaginal swabs, cervical swabs, cervicovaginal fluid, cervical biopsy specimens) at baseline and then at pre-specified timepoints after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal washing cessation (intervention) (Experimental): The intervention will consist of 3 small-group educational sessions focused on vaginal washing cessation.
  Interventions: Behavioral: Vaginal washing cessation
- Control (No Intervention): Women in the control arm will return for weekly visits (to answer study questionnaires), but will not attend group educational sessions.

INTERVENTIONS:
Behavioral: Vaginal washing cessation — Participants will attend weekly small group (~10 women per group) sessions that are structured using the transtheoretical model of behavioral change to promote vaginal washing cessation.
  Arms: Vaginal washing cessation (intervention)

SUMMARY:
Vaginal washing is a common practice that many women perceive as hygienic. However, vaginal washing has been linked to adverse reproductive health outcomes including increased HIV acquisition risk. The mechanism linking vaginal washing to HIV risk remains unknown, but may be related to increased inflammation caused by intravaginal washing practices. The primary objective of this study is to test the hypothesis that a vaginal washing cessation intervention will reduce concentrations of soluble inflammatory mediators in cervicovaginal fluid and total immune cells in mucosal tissue, reduce cervical epithelial disruption, and increase concentrations of protective vaginal Lactobacillus spp. compared to control.

DETAILED DESCRIPTION:
Vaginal washing is a common practice that many women perceive as normal and hygienic. However, vaginal washing has been linked to adverse reproductive health outcomes. Vaginal washing has been associated with increased HIV acquisition risk in a long-term open cohort study of women who engage in sex work in Mombasa, Kenya (Mombasa Cohort). Subsequent observational studies and a large individual participant data meta-analysis have supported this observation.

It has been hypothesized that the mechanism linking vaginal washing and HIV acquisition involves disruption of the vaginal microbiota. However, while some studies have demonstrated an association between vaginal washing and vaginal microbial disruption, others have not, suggesting that there may be other mechanisms linking vaginal washing and HIV acquisition risk. For example, vaginal washing could directly impact cervicovaginal inflammation, resulting in recruitment of HIV target cells and disruption of the mucosal barrier. This hypothesis is supported by preliminary findings (unpublished data) linking vaginal washing to increased concentrations of cervicovaginal IL-1 beta and a trend towards higher cervical concentrations of CD4+ T cells.

Despite the potential harms of the practice, cultural and behavioral norms may make cessation of vaginal washing difficult. To address this challenge, a pilot intervention grounded in the transtheoretical model of behavioral change for reducing vaginal washing was conducted among women in the Mombasa Cohort. After one month, all participants reported a reduction or cessation in vaginal washing practices, and at 6-12 months, 52% of women reported continued abstinence from vaginal washing. While the study was not powered to examine differences in biological outcomes related to vaginal washing, women who reduced vaginal washing during the study were observed to have fewer mucosal lesions by colposcopy, higher prevalences of cultivable Lactobacillus species (spp.), and lower concentrations of several cervicovaginal pro-inflammatory cytokines.

The primary objective of the present study is to identify the likely mechanisms linking vaginal washing and HIV acquisition risk. To achieve this objective, the investigators will conduct a randomized controlled trial of a vaginal washing cessation intervention (based in the transtheoretical model of behavioral change) to determine if a reduction in vaginal washing leads to improved mucosal homeostasis and decreased cervicovaginal inflammation by measuring i) cervicovaginal cytokine concentrations; ii) cervical immune cells from biopsy specimens; iii) expression of mucins and epithelial tight junction proteins from cervical biopsy specimens; iv) the presence of cultivable vaginal Lactobacillus spp; and, v) concentrations of select vaginal Lactobacillus spp.

ELIGIBILITY:
Inclusion Criteria:

* Reports vaginal washing beyond the introitus in the past week
* Female, aged 18-50
* Presence of a cervix
* Informed consent obtained and form signed
* HIV-seronegative
* Non-pregnant (urine β-hCG negative)
* Willing to abstain from sex for 14 days after biopsy
* Post-menarche and pre-menopause

Exclusion Criteria:

* <3 months postpartum or current breastfeeding
* Current menstruation (can enroll after menses)
* History of bleeding disorder
* Visible cervical abnormality requiring evaluation
* Medical contraindication to study protocol
* Visible cervicovaginal ulcers or lesions
* Positive test for gonorrhea, chlamydia, trichomonas, or wet preparation and examination findings indicating vulvovaginal candidiasis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Concentrations of cervicovaginal cytokines | Collected at baseline (study enrollment, time zero), at the end of the intervention (study week 4) and 3 months after enrollment (study week 12)
  Cervicovaginal cytokines will be measured from cervicovaginal fluid (collected via Softcup insertion for 15 minutes) using the Luminex platform, which is a multiplex bead-based immunoassay.
Activated CD4+ T cells and antigen presenting cells per mg cervical biopsy tissue | Collected at baseline (study enrollment, time zero), at the end of the intervention (study week 4) and 3 months after enrollment (study week 12)
  Digested cervical biopsy specimens will be stained and analyzed to detect immune cells of interest using flow cytometry
Percent cells expressing mucin or tight junction proteins | Collected at baseline (study enrollment, time zero), at the end of the intervention (study week 4) and 3 months after enrollment (study week 12)
  Expression of mucin and tight junction proteins will be detected by immunofluorescent staining of fixed cervical biopsy tissue sections and quantified
Presence of cultivable Lactobacillus spp | Collected at baseline (study enrollment, time zero), at the end of the intervention (study week 4) and 3 months after enrollment (study week 12)
  Rogosa and Columbia blood agars will be inoculated with vaginal swabs collected at study visits and the number of women with cultivable species quantified
Concentrations of Lactobacillus spp of interest | Collected at baseline (study enrollment, time zero), at the end of the intervention (study week 4) and 3 months after enrollment (study week 12)
  Concentrations of Lactobacillus spp. of interest will be measured by qPCR performed on DNA extracted from vaginal swabs collected at study visits

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sabo, Md, PhD, Principal Investigator — University of Washington